CLINICAL TRIAL: NCT02359266
Title: Clinical Trial Investigating the Role of Vitamin D in the Treatment of Depression in Patients With Chronic Liver Disease
Brief Title: Vitamin D Improves Depression in Liver Patients
Acronym: CLDVitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Dr. Caroline Stokes, Dr, Universität des Saarlandes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaarlandU
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Depression; Chronic Liver Disease
Keywords: Mood; Vitamin D deficiency; Adjuvant treatment
MeSH Terms: conditions — Depression; Vitamin D Deficiency | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D supplement (Experimental): 20,000 IU cholecalciferol p.o for the first 7 days, and weekly thereafter for 6 months
  Interventions: Dietary Supplement: Vitamin D
- Controls (No Intervention): These patients had normal vitamin D levels and did not receive any treatment with vitamin D.

INTERVENTIONS:
Dietary Supplement: Vitamin D — Given to patients with existing vitamin D deficiency
  Other Names: cholecalciferol
  Arms: Vitamin D supplement

SUMMARY:
This study evaluates the efficacy of vitamin D replacement therapy in reducing depressive symptoms in patients with chronic liver disease and vitamin D deficiency. Patients with normal vitamin D levels will be monitored as controls, and they will not receive any intervention.

DETAILED DESCRIPTION:
Patients with chronic liver diseases regularly suffer from vitamin D deficiency and depression. A recent meta-analysis reported an inverse correlation between depression and vitamin D levels. Indeed, vitamin D receptor is present and genomic and nongenomic vitamin D receptor-mediated signalling has been described in brain.

This intervention study investigates whether vitamin D therapy ameliorates depressive symptoms in chronic liver disease patients.

The investigators hypothesise that depressive symptoms will improve upon vitamin D replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* over 18 years of age
* chronic liver disease

Exclusion Criteria:

* severe hepatic encephalopathy (CFF <35 Hz)
* Interferon treatment
* hypercalcaemia (>2.7 mmol/l) or hypercalciuria (>8.0 mmol/d) with or without hyperparathyroidism (>65.0 pg/ml)
* history of calcium-containing kidney stones
* allergy or hypersensitivity to any of the supplement ingredients: peanuts, soy, gelatin
* sarcoidosis
* stage IV or V Chronic Kidney Disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes to depressive symptoms as assessed using the BDI-II score | 3 and 6 months

SECONDARY OUTCOMES:
Changes to serum liver function tests, as assessed using standard clinical-chemical assays | 3 and 6 months
Changes to bone density, as assessed using Dexa scans | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lammert, MD, Study Chair — Saarland University Medical Center; Caroline S Stokes, PhD, Principal Investigator — Saarland University Medical Center
Locations (1):
- Saarland University Medical Center, Homburg, Saarland, Germany